CLINICAL TRIAL: NCT05054686
Title: Effects of Concurrent Exercise Combinations on Pain, Function, and Proprioception in Knee Osteoarthritis: A Prospective Randomized Controlled Parallel Group Study
Brief Title: Effects of Concurrent Exercise Combinations in Knee Osteoarthritis:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda BAKTIR, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUCSEDA
Record Dates: First submitted 2021-09-12; First posted 2021-09-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: ostearthritis; pain; proprioception; resistance training; exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Parallel Group Study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination of Stretching and Aerobic Exercises at Clinic (Experimental): Combination of Stretching and Aerobic Exercises at Clinic and Strengthening and Aerobic Exercises at Home
  Interventions: Other: Stretching and Aerobic Exercise at Clinic
- Combination of Strengthening and Aerobic Exercises at Clinic (Active Comparator): Combination of Strengthening and Aerobic Exercises at Clinic and Stretching and Aerobic Exercises at Home
  Interventions: Other: Strenghthening and Aerobic Exercise
- Combination of Strengthening, Stretching and Aerobic Exercises at Clinic (Active Comparator): Combination of Strengthening, Stretching and Aerobic Exercises at Clinic and Aerobic Exercises at Home
  Interventions: Other: Strengthening, Stretching and Aerobic Exercises at clinic

INTERVENTIONS:
Other: Stretching and Aerobic Exercise at Clinic — In this group of knee osteoarthritis patients will be applied both stretching and 30 minutes bicycle exercises in the same session, strengthening exercises and 30 minutes walking will be given in seperate days as home program.
  Arms: Combination of Stretching and Aerobic Exercises at Clinic
Other: Strenghthening and Aerobic Exercise — In this group of knee osteoarthritis patients will be applied both strengthening and 30 minutes bicycle exercises in the same session, 2 days strecthing exercises and 30 minutes walking will be given in seperate days as home program.
  Arms: Combination of Strengthening and Aerobic Exercises at Clinic
Other: Strengthening, Stretching and Aerobic Exercises at clinic — In this group of knee osteoarthritis patients will be applied all stretching, strengthening and 30 minutes bicycle exercises in the same session, only 30 minutes walking will be given as home program.
  Arms: Combination of Strengthening, Stretching and Aerobic Exercises at Clinic

SUMMARY:
This study will include 3 different groups of intervention. First group of knee osteoarthritis patients will be applied both strengthening and 30 minutes bicycle exercises in the same session, 2 days strecthing exercises and 30 minutes walking will be given in seperate days as home program, Second group of knee osteoarthritis patients will be applied both stretching and 30 minutes bicycle exercises in the same session, strengthening exercises and 30 minutes walking will be given in seperate days as home program.Third group of knee osteoarthritis patients will be applied all stretching, strengthening and 30 minutes bicycle exercises in the same session, only 30 minutes walking will be given as home program. The primary outcome measures include the pain, function and the secondary outcome measures include the joint proprioception. The aim of this study is to investigate the effects on outcome measures increasing number of exercises in one session and to determine which exercise types are more suitable to prescribe as a home program.

DETAILED DESCRIPTION:
This study will include 3 different groups of intervention. First group of knee osteoarthritis patients will be applied both strengthening and bicycle exercises in the same session and strecthing exercises and walking will be given as home program in the days other than treatment session. Second group of knee osteoarthritis patients will be applied both stretching and bicycle exercises in the same session and strengthening exercises and walking will be given as home program in the days other than treatment session. Third group of knee osteoarthritis patients will be applied all stretching, strengthening and bicycle exercises in the same session and only walking exercise will be given as home program in the days other than treatment session. The primary outcome measures include the pain, function and the secondary outcome measures include the joint proprioception. The aim of this study is to investigate the effects increasing number of exercises in one session on outcome measures consisting of pain, function and proprioception. The pain will be evaluated both subjectively with numeric pain scale and WOMAC scale and objectively with pressure algometer. The function will be subjectively evaluated with WOMAC scale. The evaluation of joint proprioception will be evaluated with inclinometer. All the groups will be treated 2 days per week. The duration of total treatment lasts 8 weeks. All the groups practice aerobic exercises 2 days with bicycle ergometer application in the clinic, and 2 days walking outside as home program. Strecthing exercises will be applied for knee flexor and knee extensor muscles. Isometric strengthening exercises will be applied for knee extensor muscles. Isotonic strengthening exercises will be applied for hip extensor, flexor, abductor muscles and knee extensor and flexor muscles. The treatment outcomes will be evaluated at the end of 8 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed as knee osteoarthritis
* Being between the ages 45-74
* Being at stage 2-3 according to Kellegren Lawrence Classification
* Having body mass index lower than 30
* Being volunteer for participation to this study

Exclusion Criteria:

* Refusing to participation to study
* Having another orthopeadic problem ralated to lower extremity
* Having uncontrollable hypertension
* Having arterial and venous disease
* Having neurological disease
* Having perceptual problem
* Having cardiac pacemaker
* Participation to physiotherapy program in the last 6 months for the same extremity
* Taking injection from the same extremity in the last 6 months

Ages: 45 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index | Change of The Western Ontario and McMaster Universities Arthritis Index scores from the beginning to the end of study (8 weeks)
  The Western Ontario and McMaster Universities Arthritis Index is a questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
  Stiffness (2 items): after first waking and later in the day
  Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
  The increasing scores reflect improvement of the function.
Numeric Pain Rating Scale | Change of Numeric Pain Rating Scale scores from the beginning to the end of study (8 weeks)
  The Numeric Pain Rating Scale is a segmented numeric version of the visual analog scale in which a respondent selects a whole number (0-10 likert type integers) that best reflects the intensity of his/her pain.The levels of pain felt at rest / activity / night will be evaluated. The increase in pain scores demonstrate that the health status get worse.
Pain Pressure Treshold (PPT) | Change of Pain Pressure Treshold measurements from the beginning to the end of study (8 weeks)
  Pain Pressure Treshold is evaluated via algometric measurement that were taken from 4 point including the mid portion of patella, 3 cm medial to patellar midline, 3 cm lateral to patellar midline, 2 cm above to patellar upper boundary.The increase in algometric measurement demonstrate the development in the pain sensitivity.

SECONDARY OUTCOMES:
Proprioception | Change of Inclinometric measurements from the beginning to the end of study (8 weeks).
  Proprioception will be evaluated with digital inclinometer from 90 degree knee flexion to 30 degree knee flexion angle. The deviation from this interval reflects that the detoriation of knee joint proprioception. Therefore, decreasing deviation scores obtained from the inclinometer reflects better proprioceptive sensation.
Knee Muscle Strength | Change of muscle strength measurements from the beginning to the end of study (8 weeks)
  Muscle strength for knee flexor and extensor muscles Knee joint muscle strength was measured by using hand-held dinamometer. The measurements had taken for quadrieps and hamstring muscles. the incresing muscle strength values reflects improvement of strength of muscles around knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Seda BAKTIR, MSc.PT., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Seda Baktır, Küçükçekmece, Alkent 2000, Büyükçekmece/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We planned not to make group' data available to other researchers.